CLINICAL TRIAL: NCT05556889
Title: Safety and Analgesic Efficacy of a Modified Auriculotemporal Nerve Block: a Prospective, Randomized, Double-blind, Traditional Controlled Study
Brief Title: Safety and Analgesic Efficacy of a Modified Auriculotemporal Nerve Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Director, Principal Investigator, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ2021S195
Record Dates: First submitted 2022-03-30; First posted 2022-09-27 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Safety and Efficacy; Scalp Nerve Block
Keywords: Auriculotemporal nerve block; Scalp nerve block; safety and efficacy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- a modified auriculotemporal nerve blockade (Experimental): Helix feet in front of the zygomatic arch is served as anatomy marks of auriculotemporal nerve block, and the modified auriculotemporal nerve blockade is implemented as follows: Zygomatic arch level, posterior to the superficial temporal artery, the vertical puncture depth is about 0.5 -1 cm, and 2 ml of local anesthetics are injected after withdrawing without blood.
  Interventions: Procedure: a modified auriculotemporal nerve blockade
- Traditional auriculotemporal nerve blockade (Other): The traditional method of auriculotemporal nerve block is to inject the needle 1~1.5 cm vertically at the level of tragus and posterior of superficial temporal artery, and inject 2-3 ml of local anesthetics after pumping back without blood
  Interventions: Procedure: Traditional auriculotemporal nerve blockade

INTERVENTIONS:
Procedure: a modified auriculotemporal nerve blockade — Helix feet in front of the zygomatic arch is served as anatomy marks of auriculotemporal nerve block, and the modified auriculotemporal nerve blockade is implemented as follows: Zygomatic arch level, posterior to the superficial temporal artery, the vertical puncture depth is about 0.5 -1 cm, and 2 ml of local anesthetics are injected after withdrawing without blood.
  Arms: a modified auriculotemporal nerve blockade
Procedure: Traditional auriculotemporal nerve blockade — Traditional auriculotemporal nerve blockade
  Arms: Traditional auriculotemporal nerve blockade

SUMMARY:
1. Efficacy of a modified auriculotemporal nerve blockade for patients undergoing supratentorial craniotomy
2. Safety of a modified auriculotemporal nerve blockade for patients undergoing supratentorial craniotomy

DETAILED DESCRIPTION:
Scalp nerve block for supratentorial craniotomy patients can effectively reduce the consumption of perioperative analgesic drugs, avoid the occurrence of hypertension and tachycardia, relieve postoperative pain, improve postoperative recovery quality of patients. Scalp nerve block is safe and has fewer complications due to the small amount of local anesthetic. For auriculotemporal nerve block, temporary block of adjacent facial nerve is one of the most likely complications, with an incidence of 8.6%, and usually can be recovered within 24 hours, since the facial nerve was located in the anterior and lower part of the tragus, 1 cm deep in the skin. Therefore, improving nerve block methods and reducing the dosage of local anesthetics may reduce the risk of facial nerve block. The investigators proposed helix feet in front of the zygomatic arch as anatomy marks of auriculotemporal nerve block, and the modified auriculotemporal nerve blockade is implemented as follows: Zygomatic arch level, posterior to the superficial temporal artery, the vertical puncture depth is about 0.5 -1 cm, and 2 ml of local anesthetics are injected after withdrawing without blood. The study intends to compare a modified auriculotemporal nerve block method with the traditional way, reflecting on perioperative hemodynamical fluctuation, postoperative analgesia effect and incidence of facial nerve paralysis. This will verify the safety and analgesic efficacy of the modified nerve block method proposed in this study, and then provide a basis for improving the quality of perioperative management during neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing supratentorial craniotomy under general anesthesia;
2. 18-65 years old;
3. ASA I or II.

Exclusion Criteria:

1. Emergency surgery;
2. Be allergic to ropivacaine;
3. Participating in other clinical investigation within 30 days;
4. Skin infection at the puncture site;
5. Patients taking analgesic drugs before surgery;
6. Persons addicted to alcohol or drugs;
7. Patients with severe liver and kidney dysfunction;
8. Patients with coagulation disorder;
9. Pregnant and lactating women;
10. Patients with consciousness disorder before surgery;
11. Those who have undergone neurosurgery within the last 6 months;
12. Patients who were unable to understand the NRS before surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale (NRS) score in both groups 2 hours after surgery | 2 hours after supratentorial craniotomy
  2 hours after supratentorial craniotomy, the participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
numerical rating scale (NRS) score in both groups 8 hours after surgery | 8 hours after supratentorial craniotomy
  8 hours after supratentorial craniotomy, the participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
numerical rating scale (NRS) score in both groups 24 hours after surgery | 24 hours after supratentorial craniotomy
  24 hours after supratentorial craniotomy, the participants subjectively determine the patient's pain scores using a 0 to 10 NRS (0 = no pain; 10 = unbearable pain), to evaluate the efficacy of the modified method.
incidence of facial paralysis in both two groups | within 24 hours after supratentorial craniotomy
  within 24 hours after supratentorial craniotomy, the investigators evaluate facial nerve function of awakened participants (Diagnostic criteria for facial paralysis: unable to raise the eyebrows on the same side, unable to frown, unable to close eyes completely, or unable to smile due to facial paralysis on the same side), and record the number of patients who suffer from facial paralysis, and then calculate the incidence as: the number of patient suffering from facial paralysis/the total number in corresponding group

SECONDARY OUTCOMES:
mean arterial pressure (MAP) before anesthesia induction | before anesthesia induction
  MAP before anesthesia induction
heart rate (HR) before anesthesia induction | before anesthesia induction
  HR before anesthesia induction
MAP 3 minutes after tracheal intubation | 3 minutes after tracheal intubation
  MAP 3 minutes after tracheal intubation
HR 3 minutes after tracheal intubation | 3 minutes after tracheal intubation
  HR 3 minutes after tracheal intubation
MAP before nerve block | before nerve block
  MAP before nerve block
HR before nerve block | before nerve block
  HR before nerve block
MAP within 10 minutes after nerve block | within 10 minutes after nerve block
  MAP within 10 minutes after nerve block
HR within 10 minutes after nerve block | within 10 minutes after nerve block
  HR within 10 minutes after nerve block
MAP 1 minute after temporal region skin incision | 1 minute after temporal region skin incision
  MAP 1 minute after temporal region skin incision
HR 1 minute after temporal region skin incision | 1 minute after temporal region skin incision
  HR 1 minute after temporal region skin incision
MAP 2 minutes after temporal region skin incision | 2 minutes after temporal region skin incision
  MAP 2 minutes after temporal region skin incision
HR 2 minutes after temporal region skin incision | 2 minutes after temporal region skin incision
  HR 2 minutes after temporal region skin incision
MAP 3 minutes after temporal region skin incision | 3 minutes after temporal region skin incision
  MAP 3 minutes after temporal region skin incision
HR 3 minutes after temporal region skin incision | 3 minutes after temporal region skin incision
  HR 3 minutes after temporal region skin incision
MAP 4 minutes after temporal region skin incision | 4 minutes after temporal region skin incision
  MAP 4 minutes after temporal region skin incision
HR 4 minutes after temporal region skin incision | 4 minutes after temporal region skin incision
  HR 4 minutes after temporal region skin incision
MAP 5 minutes after temporal region skin incision | 5 minutes after temporal region skin incision
  MAP 5 minutes after temporal region skin incision
HR 5 minutes after temporal region skin incision | 5 minutes after temporal region skin incision
  HR 5 minutes after temporal region skin incision
MAP 10 minutes after temporal region skin incision | 10 minutes after temporal region skin incision
  MAP 10 minutes after temporal region skin incision
HR 10 minutes after temporal region skin incision | 10 minutes after temporal region skin incision
  HR 10 minutes after temporal region skin incision
MAP 20 minutes after temporal region skin incision | 20 minutes after temporal region skin incision
  MAP 20 minutes after temporal region skin incision
HR 20 minutes after temporal region skin incision | 20 minutes after temporal region skin incision
  HR 20 minutes after temporal region skin incision
MAP 30 minutes after temporal region skin incision | 30 minutes after temporal region skin incision
  MAP 30 minutes after temporal region skin incision
HR 30 minutes after temporal region skin incision | 30 minutes after temporal region skin incision
  HR 30 minutes after temporal region skin incision
MAP 40 minutes after temporal region skin incision | 40 minutes after temporal region skin incision
  MAP 40 minutes after temporal region skin incision
HR 40 minutes after temporal region skin incision | 40 minutes after temporal region skin incision
  HR 40 minutes after temporal region skin incision
MAP 50 minutes after temporal region skin incision | 50 minutes after temporal region skin incision
  MAP 50 minutes after temporal region skin incision
HR 50 minutes after temporal region skin incision | 50 minutes after temporal region skin incision
  HR 50 minutes after temporal region skin incision
MAP 1 hour after temporal region skin incision | 1 hour after temporal region skin incision
  MAP 1 hour after temporal region skin incision
HR 1 hour after temporal region skin incision | 1 hour after temporal region skin incision
  HR 1 hour after temporal region skin incision
MAP during surgery (at tracheal extubation) | during surgery (at tracheal extubation)
  MAP during surgery (at tracheal extubation)
HR during surgery (at tracheal extubation) | during surgery (at tracheal extubation)
  HR during surgery (at tracheal extubation)

OTHER OUTCOMES:
operation time | during surgery
  time from the time of surgery beginning until end of surgery
anesthesia time | during surgery
  time from the time of anesthesia beginning until end of anesthesia
awakening time | during surgery
  from the time of anesthesia end until time of patient awaken
PACU staying time | during surgery
  from the time coming in PACU until the time coming out PACU
anesthetic dosage | during operation
  use dosage of anesthetic drug during operation
urine volume | during operation
  urine volume during operation
bleeding volume | during operation
  bleeding volume during operation
maintenance infusion rate of remifentanil | during operation
  infusion rate of remifentanil for maintaining effective analgesic effect during operation
the dosage of remedial painkillers (remifentanil) | during operation
  the dosage of remedial painkillers (remifentanil) during operation
the dosage of remedial perdipine | during operation
  the dosage of remedial perdipine during operation
the dosage of remedial esmolol | during operation
  the dosage of remedial perdipine during operation
incidence of postoperative nausea in both two groups within 24 hours | within 24 hours after supratentorial craniotomy
  within 24 hours after supratentorial craniotomy, the investigators record the number of patients who suffer from postoperative nausea, and then calculate the incidence as: the number of patient suffering from postoperative nausea/the total number in corresponding group
incidence of postoperative vomiting in both two groups within 24 hours | within 24 hours after operation
  within 24 hours after operation, the investigators record the number of patients who suffer from postoperative vomiting, and then calculate the incidence as: the number of patient suffering from postoperative vomiting/the total number in corresponding group
incidence of hematoma at the block point in both two groups within 24 hours | within 24 hours after operation
  within 24 hours after operation, the investigators record the number of patients who suffer from hematoma at the block point, and then calculate the incidence as: the number of patient suffering from hematoma at the block point/the total number in corresponding group
incidence of infection at the block point in both two groups within 24 hours | within 24 hours after operation
  within 24 hours after operation, the investigators record the number of patients who suffer from infection at the block point, and then calculate the incidence as: the number of patient suffering from infection at the block point/the total number in corresponding group
incidence of local anesthetic toxicity in both two groups within 24 hours | within 24 hours after operation
  within 24 hours after operation, the investigators record the number of patients who suffer from local anesthetic toxicity, and then calculate the incidence as: the number of patient suffering from local anesthetic toxicity/the total number in corresponding group
the time of initial administration of remedial antiemetics within 24 hours | within 24 hours after operation
  the time of initial administration of remedial antiemetics within 24 hours after operation
the dosage of remedial antiemetics within 24 hours | within 24 hours after operation
  the dosage of remedial antiemetics within 24 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: feng gao, Principal Investigator — professor
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China